CLINICAL TRIAL: NCT02749695
Title: The Prospective, Blind, Randomized, Placebo-controlled, 4 Months Study of Efficacy of Melsmon® for Correction of Insomnia and Other Climacteric Symptoms in Premenopausal Women
Brief Title: Efficiency of Placental Drug Melsmon® in Correction of Climacteric Symptoms in Premenopausal Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Inna I. Kovalenko (Other Government)
Responsible Party: Sponsor-Investigator, Inna I. Kovalenko, Gynecologist, PhD, Resercher at the Laboratory of Gynecological Endocrinology, Scientific Center for Family Health and Human Reproduction Problems, Russia
Organization: Scientific Center for Family Health and Human Reproduction Problems, Russia (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Melsmon-913
Record Dates: First submitted 2016-04-12; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Climacteric Syndrome
Keywords: menopause, climacteric syndrome, insomnia, placental extract
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Long-Term Synaptic Depression; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Melsmon) (Experimental): 20 women used placental extract Melsmon® (Japan), 2 ml (100 mg), subcutaneously, every 2nd day for 2 weeks, then twice a week (30 injections for 4 months in total).
  Interventions: Drug: Melsmon
- Group 2 (placebo) (Placebo Comparator): 20 patients used placebo (normal saline solution): 2 ml subcutaneously, every 2nd day for 2 weeks, then twice a week (30 injections for 4 months in total).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melsmon — Placental extract Melsmon® (Japan): 2 ml (100 mg), subcutaneously, every 2nd day for 2 weeks, then twice a week (30 injections for 4 months in total).
  Other Names: Melsmon Pharmaceutical Co., Ltd.
  Arms: Group 1 (Melsmon)
Other: Placebo — 2 ml subcutaneously, every 2nd day for 2 weeks, then twice a week (30 injections for 4 months in total).
  Other Names: Normal Saline Solution
  Arms: Group 2 (placebo)

SUMMARY:
The placental drug Melsmon® is effective for correction of insomnia and other climacteric symptoms in premenopausal women. Decrease of MMI is shown both in groups with Melsmon® and Placebo, but it was more significant in patients who used Melsmon®.

DETAILED DESCRIPTION:
There were 40 women under the observation, with mild and moderate symptoms of climacteric syndrome with sleep disorders (for that the investigators evaluated modified Kupperman Index).

All patients were randomized with the help of the envelope method with the allocation ratio of 1:1 (one-to-one). 20 women were prescribed placenta extract Melsmon and 20 received placebo during 4 months.

ELIGIBILITY:
Inclusion Criteria:

* More than 40 years of age
* Irregular menstrual cycle
* Climacteric symptoms, including sleep disorders
* follicule-stimulating hormone >20 milli international units/ml -

Exclusion Criteria:

* Non-controlled hypertension (more than 140 mm Hg)
* Decompensated chronic diseases of the cardiovascular system, myocardial infarction, history of stroke
* Diabetes mellitus
* Kidney and hepatic dysfunction
* Cancer
* Breast fibroadenomas, adenomas and cysts
* Uterine fibroids with dominant nodule diameter ˃ 2 cm,
* Endometrial hyperplasia
* Individual drug idiosyncrasy
* Intake of any drugs for correction of climacteric symptoms and sleep disorders

Ages: 40 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Treatment-Related Changes of Kupperman Index | 4 months after the treatment
  kupperman index scale (score)

SECONDARY OUTCOMES:
Treatment-Related Changes of Menstrual Function | 4 months after the treatment
  ultrasound assessment of endometrium growth (mm)
Treatment-Related Changes of Depression Symptoms | 4 months after the treatment
  kupperman index questionnaire (score)
Treatment-Related Improvement in Skin Conditions | 4 months after the treatment
  the questionnaire developed by the investigators (score)
Treatment-Related Changes of Sleep Quality | 4 months after the treatment
  Pittsburgh Sleep Quality Index (score)

CONTACTS AND LOCATIONS:
Overall Officials: Larisa V. Suturina, M.D., Study Director — Scientific Center for Family Health and Human Reproduction Problems, Russia
Locations (1):
- Scientific Center for Family Health and Human Reproduction Problems, Russia, Irkutsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all available IPD: age, body mass, character of menstrual disorder and climacteric syndromes, treatment regimen (for both experimental and placebo groups), Kupperman index, results of overall-health and sleep evaluation.
  Until the publications are available, any concerned party can contact the researcher Inna I. Kovalenko (innakov2010@yandex.ru).